CLINICAL TRIAL: NCT01242098
Title: Retrospective, Real-life Observational, Matched Cohort Evaluation of the Effectiveness of BDP/FOR (Fostair® 100/6) and FP/SAL (Seretide® 125) in Patients Switching From Seretide to Fostair in UK Primary Care Asthma Management
Brief Title: Real-world Effectiveness of Combination Therapies in Primary Care Asthma Management
Acronym: Fos/Ser_switch
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Alison Chisholm, David Price, Research in Real-Life Ltd
Other Study IDs: 004/11
Record Dates: First submitted 2010-11-11; First posted 2010-11-16 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
Keywords: Asthma; Combination therapy; Primary care management; Switch; ICS/LABA; Fostair; Seretide
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fostair switch cohort: Seretide patients who, at an index date, had a step down in therapy (reduction in ICS dose of ≥50%) and switch to Fostair
  Interventions: Drug: Fixed-dose combination beclometasone dipropionate / formoterol
- Seretide continuation cohort: Seretide patients who, at an index date, had a step down in therapy (reduction in ICS dose of ≥50%) and continue on Seretide
  Interventions: Drug: Fixed dose combination salmeterol / fluticasone

INTERVENTIONS:
Drug: Fixed dose combination salmeterol / fluticasone — Branded fixed-dose combination inhaled corticosteroid / long-acting beta2-agonist therapy
  Other Names: FP/SAL; Seretide® 125
  Groups: Seretide continuation cohort
Drug: Fixed-dose combination beclometasone dipropionate / formoterol — Branded fixed-dose combination inhaled corticosteroid / long-acting beta2-agonist therapy
  Other Names: BDP/FOR; Fostair® 100/6
  Groups: Fostair switch cohort

SUMMARY:
The purpose of this study is to evaluate whether beclomethasone dipropionate / formoterol (BDP/FOR; Fostair® 100/6) is at least equivalent in terms of exacerbation prevention to fluticasone dipropionate / salmeterol (FP/SAL; Seretide® 125) in matched asthma patients switching to BDP/FOR following treatment with FP/SAL in normal clinical practice compared with patients not switched.

ELIGIBILITY:
Inclusion Criteria:

* Aged:

  * 18-60 years:
  * 61-80 years who are never-smokers
* Evidence of asthma:

  * a diagnostic code for asthma, or
  * ≥2 prescriptions for asthma at different points in time during the prior year
* Baseline FP/SAL therapy:

  * ≥2 prescription for ICS/LABA therapy as FP/SAL (Seretide® 125).

Exclusion Criteria:

* Any chronic respiratory disease other than asthma
* Are receiving maintenance oral steroid therapy during baseline period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving ICS/LABA therapy as FP/SAL (Seretide® 125) who, at an index prescription date (IPD) receive a routine asthma review* and either:
  (i) Switched to BDP/FOR (Fostair®)at same or lower BDP-equivalent ICS dose;
  OR,
  (ii) Continues on FP/SAL (Seretide® 125) for the duration of the outcome period at the same or lower BDP-equivalent ICS dose prescribed at baseline.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate | One-year outcome period
  Where an exacerbation is defined as:
  (i) Asthma-related
  1. Hospital attendance / admissions OR
  2. Accident & Emergency (A&E) attendance OR
  (ii) Use of oral steroids.

SECONDARY OUTCOMES:
Exacerbation control (a composite proxy measure) | One-year outcome period
  Controlled:
  Absence of:
  (i) Asthma-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours consultations, OR
  4. Out-patient department attendance
  (ii) GP consultations for lower respiratory tract infection
  (iii) Prescriptions for acute courses of oral steroids
Treatment success 1 | One-year outcome period
  (i) Exacerbation control
  AND
  (ii) No change in therapeutic regimen:
  * ≥50% increase in ICS dose relative to IPD dose, and/or
  * Change in ICS/LABA drug within class, and/or
  * Change in delivery device, and/or
  * Use of additional (defined as not received during baseline year) therapy as defined by: theophylline, leukotriene receptor antagonists (LTRAs).
Asthma hospitalisations | One-year outcome period
  1. Definite: Hospitalisations coded with an asthma read code
  2. Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of an asthma read code
Compliance with ICS/LABA therapy | One-year outcome period
  Compliance calculation based on prescription refills and (where possible) compliance questionnaire data
Use of reliever medication | One-year outcome period
  average daily dosage during outcome year. Outcome SABA usage will be categorised within ranges used to match baseline SABA use to optimise matching of the treatment arms.
Cost of therapeutic regimen. | One-year outcome period
  Mean healthcare costs (drug costs + consultation, admission costs, etc - total and respiratory-related) per patient recorded during the outcome year
Asthma-related / respiratory hospitalisations | one year outcome period
  1. Definite: Hospitalisations coded with a lower respiratory code
  2. Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of a lower respiratory read code
Oral Thrush | One-year outcome period
  Identified as:
  (i) Topical oral anti-fungal prescriptions, and / or
  (ii) Coded for oral candidiasis

CONTACTS AND LOCATIONS:
Locations (1):
- Optimum Patient Care, Cawston, Norfolk, United Kingdom

REFERENCES:
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org